CLINICAL TRIAL: NCT01719068
Title: Early Detection of Lung Cancer and Mesothelioma in Workers Exposed to Asbestos
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: BC Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: H12-01812
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Mesothelioma; Lung Cancer
Keywords: Mesothelioma; Lung Cancer; Early Detection
MeSH Terms: conditions — Mesothelioma; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Workers exposed to asbestos

SUMMARY:
This is a pilot study that aims to develop a lung cancer screening program for workers in British Columbia, Canada exposed to asbestos who are at risk of developing lung cancer/pleural mesothelioma. This is high risk population is at of respiratory system diseases as a result of their occupational exposures. Additionally, knowledge garnered from this study will allow us to develop other studies that will further our understanding of asbestos related lung cancer and mesothelioma.

ELIGIBILITY:
Inclusion Criteria:

* Women or men age 50 to 79 years
* history of exposure to asbestos at work and one or more of the following:

  * lung cancer risk ≥2% over 3 years or
  * asbestosis or pleural plaques on a chest x-ray or
  * abnormal auto-antibodies level using the EarlyCDT test
* Capable of providing informed consent for screening procedures (low dose spiral CT, lung function, blood biomarkers).

Exclusion Criteria:

* Any medical condition, such as severe heart disease (e.g. unstable angina, chronic congestive heart failure), acute or chronic respiratory failure, or any disorder, that in the opinion of the physician unlikely to benefit from screening due to shortened life-expectancy from co-existing illnesses
* Have been previously diagnosed with mesothelioma
* Have had other cancer within the past 5 years with the exception of the following cancers: non-melanomatous skin cancer,localized prostate cancer, carcinoma in situ (CIS) of the cervix, or superficial bladder cancer. Treatment of the exceptions must have ended >6 months before registration into this study
* Pregnancy
* Unwilling to have a low dose CT scan of chest
* Unwilling to sign a consent

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Workers in British Columbia who have been exposed to asbestos.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Development of Model to Predict Workers at highest risk of lung cancer/mesothelioma | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lam, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- British Columbia Cancer Agency, Vancouver, British Columbia, Canada